CLINICAL TRIAL: NCT06741319
Title: The Institute of HIV Research and Innovation (IHRI)
Brief Title: Behavioral and Psychosocial Characteristics of Clients Accessing Services at IHRI
Status: Recruiting | Type: Observational
Sponsor: Institute of HIV Research and Innovation Foundation, Thailand (Other)
Responsible Party: Sponsor
Other Study IDs: IHRI009
Record Dates: First submitted 2024-12-12; First posted 2024-12-18 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: HIV
MeSH Terms: interventions — Sex; Referral and Consultation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Demographic characteristics — * Gender identity
  * Sex assigned at birth
  * Age
  * Address
  * History of study enrollment(s)
Behavioral: Social and sexual behaviors — * Places where clients go for shopping, dining out, exercise, entertainment
  * Places where clients meet their sexual partner(s)
  * Places where clients obtain condoms and lubricants
  * Social networking and other online services clients regularly use and purposes of using
  * Lifetime and current sexual practices and condom use
  * Number and types of sexual partners
  * Self-perceived HIV risk level
  * Disclosure of HIV or sexual orientation status
Behavioral: Psychosocial characteristics — * Sexual orientation
  * Educational level
  * Occupation and income
  * Attitude towards and use of HIV testing and sexual health services
  * Use of injecting drugs, recreational drugs, and alcohol
Behavioral: Clinical characteristics — * Medical history, including gender dysphoria and hormone therapy
  * HIV counseling and testing
  * Diagnosis and treatment of sexually transmitted diseases (STD)
  * Sample collection information
  * Laboratory results
  * Gender dysphoria and mental health history
  * Body hair pattern
  * Bridging therapy
  * Fertility and reproductive issues
  * Gender transition effects
Behavioral: Referral and linkage to care for HIV-positive clients — * Health insurance scheme
  * Initiation and continuation of antiretroviral treatment
Behavioral: Characteristics associated with service implementation — - Facilitators, barriers, feasibility and acceptability of and satisfaction with service implementation as identified by clients and healthcare providers

SUMMARY:
This protocol describes a 20-year prospective cohort study, gathering behavioral and psychosocial information on clients who access services of the Institute of HIV Research and Innovation (IHRI) and the Thai Red Cross AIDS Research Centre through the Thai Red Cross Anonymous Clinic, the Thai Red Cross Mobile Clinics, Affiliated Health Clinics, The gender and immunity clinic and Pribta Tangerine Polyclinic. Services provided through these sites include VCT, STD screening and treatment, anal and cervical Pap smears, general health checkups, sexual health education, and sexual health communication, gender-affirmative hormone therapy (GAHT) and risk-reduction via web boards and chat rooms.

Behavioral and psychosocial information will be collected using validated questionnaires and from data collection forms routinely used when providing services in different service sites of IHRI and the TRC-ARC. The information will be collected anonymously at baseline and at follow-up visits, according to type of services each client receives. Clients at the Thai Red Cross Anonymous Clinic, Thai Red Cross Mobile Health Clinics, Affiliated Health Clinics and Pribta Tangerine Polyclinic will be given an identification number.

Qualitative methods, including focus group discussions (FGD) and in-depth interviews (IDI) will be conducted with clients and healthcare providers to examine the facilitators, barriers, feasibility and acceptability of service implementation.

DETAILED DESCRIPTION:
STUDY OBJECTIVES

1. To describe behavioral and psychosocial characteristics of clients who access services.
2. To understand the effectiveness of the HIV prevention package offered to clients who access services in terms of cost and infections averted
3. To study changes in behavioral and psychosocial characteristics among clients over time
4. To study differences in behavioral and psychosocial characteristics among clients by gender identity, sexual orientation, HIV status, and service sites
5. To assess behavioral and psychosocial factors that influence the willingness to participate in study trials
6. To assess the facilitators, barriers, feasibility and acceptability of and satisfaction with service implementation among clients and healthcare providers under IHRI and TRCARC

ELIGIBILITY:
Inclusion Criteria:

1. 18 years or 16 and 17 years of age with parental or guardian consent In non- or pre-SRS cases
2. Recommendation1 by counsellor based on:

   A) Presence of GD history B) Understanding of risks and benefits of GAHT D) Practice and readiness for gender transition E) Availability of social support F) Ability to take hormones as instructed
3. Verbal informed consent or signed informed consent on file
4. No exclusionary medical conditions
5. Approved by physician

In SRS- and post-SRS cases2

1. Verbal informed consent or signed informed consent on file
2. No exclusionary medical conditions
3. Approved by physician

Exclusion Criteria:

None

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Study population: Clients accessing services of the Pribta Tangerine Polyclinic, the Thai Red Cross Anonymous Clinic, the Thai Red Cross Mobile Clinics and Affiliated Health Clinics.
Sampling Method: Probability Sample
Enrollment: 300000 (Estimated)
Dates: Start 2013-07-02 (Actual); Primary Completion 2027-07-02 (Estimated); Study Completion 2030-07-02 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome Measure | 20 years
  1. Demographic characteristics
  2. Social and sexual behaviors
  3. Psychosocial characteristics
  4. Clinical characteristics
  5. Referral and linkage to care for HIV-positive clients
  6. Characteristics associated with service implementation

CONTACTS AND LOCATIONS:
Overall Officials: Siriporn Nonenoy, BNH,MPH, Study Chair — Institute of HIV Research and Innovation
Locations (1):
- Tangerine Clinic, Institute of HIV Research and Innovation, Pathum Wan, Bangkok, Thailand